CLINICAL TRIAL: NCT05085366
Title: A Phase 3, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of mRNA-1647 Cytomegalovirus (CMV) Vaccine in Healthy Participants 16 to 40 Years of Age
Brief Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of mRNA-1647 Cytomegalovirus (CMV) Vaccine in Healthy Participants 16 to 40 Years of Age
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor decided to terminate the study after it did not meet the primary efficacy endpoint at final analysis. The safety profile was consistent with prior studies, and no safety concerns were raised by the Data and Safety Monitoring Board.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1647-P301; 2020-006051-17 (EudraCT Number); 2023-508820-37-00 (Other: EU CTR Number)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cytomegalovirus Infection
Keywords: mRNA-1647; Moderna; Cytomegalovirus; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Congenital; Virus Diseases; Infection Viral; DNA Virus Infections; Messenger RNA
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases; DNA Virus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1647 (Experimental): Participants will receive mRNA-1647 vaccine by intramuscular (IM) injection on Day 1, Day 57, and Day 169.
  Interventions: Biological: mRNA-1647
- Placebo (Placebo Comparator): Participants will receive mRNA-1647 vaccine matching placebo by IM injection on Day 1, Day 57, and Day 169.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Lyophilized product that is reconstituted with 0.9% sodium chloride (normal saline)
  Arms: mRNA-1647
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of mRNA 1647 vaccine in CMV-seronegative female participants and to evaluate the safety and reactogenicity of mRNA-1647 vaccine in all participants. The purpose of the Phase 3 extension substudy is to extend the observation period of the main study and to assess the longer-term immunogenicity, efficacy, and safety of the mRNA-1647 vaccine against primary CMV infection in healthy females who were CMV-seronegative at Baseline of the mRNA-1647-P301 main study (including participants who remain CMV-seronegative upon entry into the extension substudy and participants who seroconverted during the main study). The extension substudy will also evaluate the immune persistence and safety of mRNA-1647 in a subset of female participants who were CMV-seropositive at Baseline of the main study. No interventional vaccine will be administered in the extension substudy.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants aged ≥20 years, has or anticipates having direct exposure within 7 months after the planned first dose (in the home, socially, or occupationally) to at least 1 child ≤5 years of age. Direct exposure is defined as either participant is the parent, or participant has close contact (feeding, diaper changes, childcare/supervision) for at least 8 hours per week.
* CMV-seronegative Cohort is CMV-seronegative based on CMV testing at Screening.
* CMV-seropositive Cohort is CMV-seropositive based on CMV testing at Screening.
* Investigator assessment confirms that the participant (including in the case of an emancipated minor), or parent(s)/legally acceptable representative (LAR)(s), as applicable, understand and are willing and physically able to comply with protocol-mandated follow-up including all study visits and procedures anticipated during the 30 month study period.
* Female participants of child-bearing potential: Urine pregnancy test is negative at Screening and negative on the day of the first injection (Day 1). If the participant is sexually active with men, has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection (Day 1) and agrees to continue adequate contraception through 3 months following the third study injection (Month 9/Day 257).

Extension substudy:

* All consenting participants who were CMV-seronegative at Baseline in the mRNA-1647-P301 main study (including those who did seroconvert and did not seroconvert during the main study), received at least one study injection in the main study but did not withdraw study consent, and completed the final study visit in mRNA-1647-P301 main study.
* Consenting participants in mRNA-1647-P301 main study who were CMV-seropositive at Baseline, received all 3 study injections, did not withdraw study consent, and completed the final study visit in the main study.

Key Exclusion Criteria:

* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Received or plans to receive any nonstudy vaccine <28 days prior to and after any study injection; in addition, the following criteria for COVID-19 and influenza vaccines apply:
* Any COVID-19 primary vaccination series must have been completed a minimum 28 days prior to receiving any dose of the study injection.
* COVID-19 vaccines (including any booster dose, regardless of manufacturer) must be administered at least 28 days prior to or after any study injection.
* Influenza vaccines may be administered > 14 days prior to or after any study injection.
* Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the day of first injection (Day 1) (for corticosteroids, ≥5 milligrams (mg)/day of prednisone equivalent) or plans to do so during the course of the study. Inhaled, nasal, and topical steroids are allowed. Stable immunomodulator regimens used for managing environmental allergies are allowed.
* Receipt of an antiviral with activity against CMV (ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir, acyclovir, valacyclovir) <2 weeks prior to the day of first injection or plans to do so during the course of the study.
* Previous receipt of an investigational CMV vaccine.
* Receipt of systemic immunoglobulins or blood products <3 months prior to the day of first injection.
* Participated in an interventional clinical study <28 days prior to the day of first injection (Day 1) or plans to do so while enrolled in this study.
* Participant has donated ≥450 milliliters (mL) of blood products <28 days prior to Screening.
* Participant is a member of study team or is an immediate family member or household member of study personnel.

Extension substudy:

* Receipt of any CMV vaccine other than mRNA-1647.
* Diagnosis or condition that, in the judgment of the Investigator, may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures, including any medical, psychiatric, or occupational condition that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7454 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Seroconversion From a Negative to a Positive Result for Serum Immunoglobulin G (IgG) Against Antigens not Encoded by mRNA-1647 | Day 197 (28 days after the third injection) up to Day 887 (24 months after the third injection)
Number of Participants With Solicited Adverse Reactions (ARs) | Up to 176 days (7 days after each injection)
Number of Participants With Unsolicited Adverse Events (AEs) | Up to 197 days (28 days after each injection)
Number of Participants With Medically-Attended Adverse Events (MAAEs) | Day 1 through 6 months after the last injection (up to 347 days)
Number of Participants With Adverse Event of Special Interests (AESIs) and Serious Adverse Events (SAEs) | Day 1 through Month 30
Geometric Mean Titers (GMTs) of Antigen-Specific Neutralizing Antibody (nAb) | Month 30 up to Month 54
Geometric Mean Concentration (GMC) of Binding Antibody | Month 30 up to Month 54
Seroconversion From a Negative to a Positive Result for Serum IgG Against Antigens not Encoded by mRNA-1647 | Month 30 up to Month 54
Number of Participants With Systemic Viral Dissemination | Month 30 up to Month 54

SECONDARY OUTCOMES:
GMTs of Antigen-Specific nAb | Day 1, Months 3, 7, 12, 18, 24, and 30
GMC of Antigen-Specific Binding Antibody | Day 1, Months 3, 7, 12, 18, 24, and 30
Number of Participants with AEs leading to Study Discontinuation, SAEs and Deaths | Month 30 up to Month 54
Number of Participants With Systemic Viral Dissemination | Day 1 through Month 30
Number of Participants With Positive Urine CMV Polymerase Chain Reaction (PCR) Results Post Seroconversion | Day 1 through Month 30
Number of Participants With Positive Urine CMV PCR Results Post Seroconversion | Month 30 up to Month 54

CONTACTS AND LOCATIONS:
Locations (293):
- United States (180):
  - Central Research Associates Inc, Birmingham, Alabama
  - Accel Research Site - Achieve - Birmingham - ERN - PPDS, Birmingham, Alabama
  - SEC Clinical Research LLC - Dothan - ClinEdge - PPDS, Dothan, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Chandler Clinical Trials, LLC, Chandler, Arizona
  - Arizona Clinical Trials, Mesa, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - Hope Research Institute LLC, Phoenix, Arizona
  - Epic Medical Research Arizona, Surprise, Arizona
  - Voyage Medical, Tempe, Arizona
  - Hope Research Institute LLC, Tempe, Arizona
  - Tucson Neuroscience Research - M3 WR - ERN - PPDS, Tucson, Arizona
  - The Institute for Liver Health-Tucson, Tucson, Arizona
  - Del Sol Research Management - ClinEdge - PPDS, Tucson, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - Applied Research Center of Arkansas - Clinedge - PPDS, Little Rock, Arkansas
  - Velocity Clinical Research - Banning, Banning, California
  - Velocity Clinical Research - Chula Vista, Chula Vista, California
  - Apex Research Group, Fair Oaks, California
  - Ascada Research LLC, Fullerton, California
  - Paradigm Clinical Research Center, La Mesa, California
  - Velocity Clinical Research - San Diego, La Mesa, California
  - Long Beach Research Institute, LLC, Long Beach, California
  - Long Beach Clinical Trials Services Inc., Long Beach, California
  - Catalina Research Institute LLC, Montclair, California
  - Carbon Health- NoHo West Urgent Care and Primary Care, North Hollywood, California
  - Empire Clinical Research, Pomona, California
  - Paradigm Clinical Research Institute, Inc. - ClinEdge, Redding, California
  - Smart Cures Clinical Research, Rolling Hills Estates, California
  - Northern California Research Corp, Sacramento, California
  - Womens Healthcare Research Corporation ERN PPDS, San Diego, California
  - Care Access Research - Santa Clarita, Santa Clarita, California
  - Stanford University School of Medicine, Stanford, California
  - Clinical Trials Management Services, LLC, Thousand Oaks, California
  - Bayview Research Group, Valley Village, California
  - Next Level Clinical Trials, West Covina, California
  - Care Access Research - Aurora, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Paradigm Clinical Research Institute Inc - ClinEdge, Wheat Ridge, Colorado
  - New England Research Associates LLC - ERN - PPDS, Bridgeport, Connecticut
  - Clinical Research Consultants LLC, Milford, Connecticut
  - Emerson Clinical Research Institute LLC - Kennedy St, Washington D.C., District of Columbia
  - Invictus Clinical Research Group, LLC, Coconut Creek, Florida
  - Luna Research LLC, Coral Gables, Florida
  - Herco Medical and Research Center, Inc., Coral Gables, Florida
  - Precision Clinical Research, LLC, Coral Springs, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Unique Clinical Trials, LLC, Doral, Florida
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Best Quality Research, Inc, Hialeah, Florida
  - Florida International Medical Research, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Spotlight Research Center, LLC, Miami, Florida
  - Floridian Clinical Research - ClinEdge - PPDS, Miami Lakes, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Emerald Coast OBGYN Clinical Research, Panama City, Florida
  - Ideal Clinical Research, Inc. - ClinEdge - PPDS, Pembroke Pines, Florida
  - Precision Clinical Research - Plantation, Plantation, Florida
  - GCP Global Clinical Professionals, St. Petersburg, Florida
  - Tampa Bay Health Care, Tampa, Florida
  - CVS HealthHub - Atlanta S, Atlanta, Georgia
  - CVS HealthHub - Atlanta, Atlanta, Georgia
  - Tekton Research - Georgia - Platinum, Chamblee, Georgia
  - Centricity Research - Roswel, Columbus, Georgia
  - CVS HealthHub - Dacula, Dacula, Georgia
  - IResearch Atlanta LLC, Decatur, Georgia
  - CVS HealthHub - Kennesaw, Kennesaw, Georgia
  - Drug Studies America - ClinEdge - PPDS, Marietta, Georgia
  - CVS HealthHub - Mcdonough, McDonough, Georgia
  - CVS HealthHub - Newman, Newnan, Georgia
  - One Health Research Clinic, Inc., Norcross, Georgia
  - Mount Vernon Clinical Research, LLC - M3 WR - ERN - PPDS, Sandy Springs, Georgia
  - CVS HealthHub - Savannah, Savannah, Georgia
  - Clinical Research Prime - Clinedge, Idaho Falls, Idaho
  - Velocity Clinical Research, Meridian, Idaho
  - Affinity Health, Oak Brook, Illinois
  - Optimal Research, Peoria, Illinois
  - ASHA Clinical Research - ClinEdge, Hammond, Indiana
  - Del Pilar Medical and Urgent Care, Mishawaka, Indiana
  - Iowa Clinic, Des Moines, Iowa
  - Johnson Country Clin-Trials, Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Velocity Clinical Research - Covington, Metairie, Louisiana
  - Centennial Medical Group - Elkridge - Rx Trials, Elkridge, Maryland
  - Meridian Clinical Research-(Rockville Maryland), Rockville, Maryland
  - DM Clinical Research - The Brook House, Brookline, Massachusetts
  - Skylight Health Research - Burlington, Burlington, Massachusetts
  - ActivMed Practices & Research Inc, Methuen, Massachusetts
  - Voyage Medical - Michigan, Canton, Michigan
  - Wayne State University, Detroit, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research - Southfield, Southfield, Michigan
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - University of Minnesota Clinical Research Unit, Minneapolis, Minnesota
  - MedPharmics, LLC, Gulfport, Mississippi
  - MediSync Clinical Research Hattiesburg Clinic, Petal, Mississippi
  - Boeson Research GTF - Great Falls, Great Falls, Montana
  - Boeson Research KAL - Kalispell - ERN - PPDS, Kalispell, Montana
  - Boeson Research MSO - Missoula, Missoula, Montana
  - Meridian Clinical Research (Grand Island, Nebraska), Grand Island, Nebraska
  - Meridian Clinical Research (Hastings, Nebraska), Hastings, Nebraska
  - Be Well Clinical Studies, LLC - Lincoln - ERN - PPDS, Lincoln, Nebraska
  - Meridian Clinical Research (Norfolk-Nebraska), Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research-(Omaha Nebraska), Omaha, Nebraska
  - Clinical Research Center Of Nevada, Las Vegas, Nevada
  - Med Clinic Research Partners, LLC, Irvington, New Jersey
  - Albuquerque Clinical Trials Inc., Albuquerque, New Mexico
  - MedPharmics, LLC. - Albuquerque, Albuquerque, New Mexico
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Binghamton, New York
  - WellNow Urgent Care Clinical Research, East Amherst, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Carolina Institute for Clinical Research - M3 WR - ERN - PPDS, Fayetteville, North Carolina
  - Monroe Biomedical Research (Venus St), Monroe, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - M3 Wake Research, Inc - M3 WR - ERN - PPDS, Raleigh, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - CTI Clinical Research Center - ClinEdge - PPDS, Cincinnati, Ohio
  - Meridian Cincinnati, Cincinnati, Ohio
  - University of Cincinnati Medical Center-Goodman St, Cincinnati, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - WellNow Urgent Care & Research - Huber Heights, Columbus, Ohio
  - PriMed Clinical Research - ClinEdge, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Epic Medical Research Oklahoma, Chickasha, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tekton Research - Oklahoma - Platinum, Yukon, Oklahoma
  - Velocity Clinical Research - Medford, Medford, Oregon
  - SPICA Clinical Research, Columbia, South Carolina
  - PMG Research of Charleston LLC, Mt. Pleasant, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - Premier Family Physicians - Austin - Hunt, Austin, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Gadolin Research LLC, Beaumont, Texas
  - REX Clinical Trials, Beaumont, Texas
  - Tekton Research - Beaumont, Beaumont, Texas
  - Velocity Clinical Research - Austin, Cedar Park, Texas
  - Global Medical Research, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - ANRC Research, El Paso, Texas
  - Village Health Partners Frisco Medical Village, Frisco, Texas
  - Trio Clinical Trials LLC, Houston, Texas
  - Vilo Research Group, L.L.C., Houston, Texas
  - New Horizon Medical Group, LLC, Houston, Texas
  - Cedar Health Research - Fort Worth - PPDS, Irving, Texas
  - Helios CCR, Inc.-keller-PPDS, Keller, Texas
  - University of Texas Medical Branch - Bay Colony, SIVS Clinical Trials Program, League City, Texas
  - BRCR Medical Center Inc - McAllen, McAllen, Texas
  - Synergy Group US, LLC, Missouri City, Texas
  - Austin Regional Clinic ARC Clinical Research at Kelly Lane, Pflugerville, Texas
  - GLRI McAllen Research, Pharr, Texas
  - ACRC Trials - Independence Parkway - Plano - Hunt - PPDS, Plano, Texas
  - Epic Medical Research LLC, Red Oak, Texas
  - Clinical Trials of Texas, Inc. - HyperCor, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Crossroads Clinical Research (Victoria), Victoria, Texas
  - ClinPoint Trials LLC, Waxahachie, Texas
  - Tanner Clinic, Layton, Utah
  - Granger Medical Clinic - Riverton, Riverton, Utah
  - Foothill Family Clinic, Salt Lake City, Utah
  - Foothill Family Clinic - South Clinic, Salt Lake City, Utah
  - Velocity Clinical Research, West Jordan, Utah
  - Health Research of Hampton Roads Inc. - ClinEdge, Newport News, Virginia
  - York Clinical Research, Norfolk, Virginia
  - David Ramstad Associates Research - IACT - HyperCore - PPDS, Suffolk, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Seattle Clinical Research Center, Seattle, Washington
  - Velocity Clinical Research - Spokane - PPDS, Spokane, Washington
  - University Of Wisconsin - Madison, Madison, Wisconsin
- Australia (15):
  - Paratus Clinical Research, Bruce, Australian Capital Territory
  - Paratus Clinical Research - Western Sydney, Blacktown, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Northside Health, Coffs Harbour, New South Wales
  - Kanwal Medical Complex, Kanwal, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Emeritus Research, Botany, North South Wales
  - University of the Sunshine Coast, Health Hub Morayfield, Morayfield, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - USC Southbank, Southbank, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
  - The University of Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Telethon Kids Institute, Nedlands, Western Australia
- Belgium (3):
  - Center for Vaccinology (CEVAC), Ghent, Oost-Vlaanderen
  - AZ Sint-Lucas Brugge, Bruges, West-Vlaanderen
  - CHU de Liège, Liège
- Canada (16):
  - University of Alberta Hospital, Edmonton, Alberta
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - LMC Manna Research - Burlington - HyperCore - PPDS, Burlington, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Centricity Research - Toronto, Toronto, Ontario
  - Centricity Research - Quebec - HyperCore - PPDS, Lévis, Quebec
  - Centricity Research - Mirabel - HyperCore - PPDS, Mirabel, Quebec
  - McGill University Health Center, Montreal, Quebec
  - McGill University Health Centre-Vaccine Study Centre, Pierrefonds, Quebec
  - Centricity Research - Montreal - HyperCore - PPDS, Pointe-Claire, Quebec
  - Diex Recherche - Québec - HyperCore, Québec, Quebec
  - Diex Recherche - Joilette - HyperCore - PPDS, Saint-Charles-Borromée, Quebec
  - Diex Recherche - Sherbrooke - HyperCore, Sherbrooke, Quebec
  - Diex Recherche - Victoriaville - HyperCore, Victoriaville, Quebec
- Estonia (5):
  - CCBR Clinical Research, Tallinn, Harju
  - Al Mare Family Doctors Centre, Tallinn, Harju
  - Merelahe Family Doctors Centre, Tallinn, Harju
  - Vee Family Doctors Center Ltd, Paide, Järvamaa
  - Clinical Research Centre Ltd., Tartu, Tartu
- Finland (10):
  - Etelä Helsingin Rokotetutkimusklinikka, Helsinki, Etelä-Suomen Lään
  - Kokkolan Rokotetutkimusklinikka, Kokkola, Keski-Pohjanmaa
  - Oulun Rokotetutkimusklinikka, Oulu, Oulun Lääni
  - Tampereen Rokotetutkimusklinikka, Tampere, Pirkanmaa
  - Porin Rokotetutkimusklinikka, Pori, Satakunta
  - Tampereen Yliopisto Seinajoen Rokotusklinikka, Seinäjoki, South Ostrobothnia
  - Espoon rokotetutkimusklinikka, Espoo, Uusimaa
  - Itä Helsingin Rokotetutkimusklinikka, Helsinki, Uusimaa
  - Järvenpään Rokotetutkimusklinikka, Jarvenpaa, Uusimaa
  - Turun Rokotetutkimusklinikka, Turku, Västra Finlands Län
- France (9):
  - CHRU Nantes, Nantes, Pays de la Loire Region
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier et Universitaire de Limoges, Limoges
  - CHU Montpellier - Hôpital St Eloi, Montpellier
  - Hopital Necker, Paris
  - Groupe Hospitalier Cochin Saint Vincent de Paul, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - CHRU de Tours, Tours
- Germany (15):
  - TriDerm, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Frauenarztpraxis Erwin Göckeler-Leopold, Geseke, North Rhine-Westphalia
  - Dermatologie Quist, Mainz, Rhineland-Palatinate
  - Klifeck GmbH, Delitzsch, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Praxis Reinfeld-Mitte, Reinfeld, Schleswig-Holstein
  - Berliner Centrum für Reise- und Tropenmedizin BCRT GmbH, Berlin
  - Bernhard Nocht Centre for Clinical Trials (BNCCT)am Bernhard-Nocht-Institut für Tropenmedizin, Hamburg
  - Velocity Clinical Research - Hamburg - PPDS, Hamburg
  - Office of Klaus H. Peters, Dr.med, Hamburg
  - Velocity Clniical Research Leipzip Gmbh, Leipzig
  - AmBeNet GmbH, Leipzig
  - Centrum Für Diagnostik und Gesundheit, München
  - Medislim GmbH - Zentrum fuer Ambulante Klinische Forschung, Weinheim
- Israel (10):
  - Sheba Medical Center - PPDS, Petah Tikva, Central District of Israel
  - Rambam Medical Center - PPDS, Haifa, Haifa Hefa
  - Shamir Medical Center Assaf Harofeh, Beer Yaakov, Rishon Lezion
  - Soroka University Medical Centre, Beer Sheva, Tel Aviv
  - Maccabi Hashalom, Tel Aviv, Tel Aviv
  - Hadassah Medical Center - PPDS, Jerusalem, Yerushalayim Al Quds
  - Shaare Zedek Medical Center, Jerusalem, Yerushalayim Al Quds
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (2):
  - Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS San Gerardo dei Tintori - MBBM - c/o Centro Maria Letizia Verga, Monza
- Japan (13):
  - Clinical Trial Site, Funabashi-shi, Chiba
  - Clinical trial site, Fukuoka, Fukuoka
  - Clinical Trial Site, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyôgo
  - Clinical trial site, Osaka-shi Osaka, Kansai
  - Clinical Trial Site, Habikino-shi, Osaka
  - Clinical Trial Site, Osaka, Osaka
  - Clinical Trial Site, Sakai-shi, Osaka
  - Clinical Trial Site, Kawagoe-shi, Saitama
  - Clinical Trial Site, Chuo-ku, Tokyo
  - Clinical Trial Site, Shibuya-ku, Tokyo
  - Clinical Trial Site, Shinjuku, Tokyo
  - Clinical Trial Site, Taito-ku, Tokyo
- Spain (8):
  - C.H. Regional Reina Sofia, Córdoba, Andalusia
  - Hospital Quironsalud Malaga, Málaga, Andalusia
  - Instituto Hispalense de Pediatria, Seville, Andalusia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - ABS Centelles, Centelles, Catalonia
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela, Galicia
  - Hospital HM Puerta del Sur, Móstoles, Madrird
  - Hospital Universitario La Paz., Madrid
- United Kingdom (7):
  - The James Cook University Hospital, Middlesbrough, Cleveland
  - William Harvey Clinical Research Centre, London, England
  - St George s Vaccine Institute, London, England
  - Lakeside Surgery, Corby, Northamptonshire
  - NIHR Patient Recruitment Centre: Newcastle, Newcastle upon Tyne, Northumberland
  - St Michaels Hospital, Bristol, South West England
  - NIHR Clinical Research Facility, University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Galiza EP, Khalil A, Heath PT. Update on Vaccines in Antenatal Care. Pediatr Infect Dis J. 2024 Feb 1;43(2):e60-e62. doi: 10.1097/INF.0000000000004183. Epub 2023 Dec 27. No abstract available. PMID 38190492
- [Derived] Stewart AG, Kotton CN. What's New: Updates on Cytomegalovirus in Solid Organ Transplantation. Transplantation. 2024 Apr 1;108(4):884-897. doi: 10.1097/TP.0000000000004855. Epub 2023 Oct 30. PMID 37899366
- [Derived] Kadambari S, Evans C, Lyall H. Congenital Infections: Priorities and Possibilities for Resource-limited Settings. Pediatr Infect Dis J. 2023 Feb 1;42(2):e45-e47. doi: 10.1097/INF.0000000000003710. Epub 2022 Sep 12. No abstract available. PMID 36102707